CLINICAL TRIAL: NCT03027180
Title: DIFFERENT LEVELS OF NONINVASIVE POSITIVE AIRWAY PRESSURE FOR LUNG EXPANSION ON PATIENTS WITH PLEURAL DRAINAGE: A STUDY VIA COMPUTED TOMOGRAPHY
Brief Title: Pressure Levels on Lung Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Adriana Claudia Lunardi, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UNICID/CNPq 442709/2014-5
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0 (zero) cmH2O (Active Comparator): After draining, people will be asked about the level of pain via visual numeric scale and then subjected to chest computed tomography (Aquilion 64-Toshiba Medical Systems®, Japan), using positive airway pressure in the airways with 0 cmH2O
  Interventions: Device: Noninvasive positive airway pressure with different levels
- 4 cmH2O (Experimental): After draining, people will be asked about the level of pain via visual numeric scale and then subjected to chest computed tomography (Aquilion 64-Toshiba Medical Systems®, Japan), using positive airway pressure in the airways with 4 cmH2O
  Interventions: Device: Noninvasive positive airway pressure with different levels
- 15 cmH2O (Experimental): After draining, people will be asked about the level of pain via visual numeric scale and then subjected to chest computed tomography (Aquilion 64-Toshiba Medical Systems®, Japan), using positive airway pressure in the airways with 15 cmH2O
  Interventions: Device: Noninvasive positive airway pressure with different levels

INTERVENTIONS:
Device: Noninvasive positive airway pressure with different levels

SUMMARY:
Question: What level of noninvasive positive airway pressure is able to expand the lungs of people with pleural drainage? Design: Cross-sectional, experimental and randomized study. Participants: Four consecutive people with pleural effusion drained within 24 hours, with controlled pain and without contraindications to use of noninvasive positive pressure. Intervention: Each person will be randomly subjected to three levels of noninvasive positive airway pressure: 0 (zero), 4 and 15 cmH2O for evaluation via chest computed tomography. Outcome measures: Lung area.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* presence of pleural drainage after traumatic hemothorax
* thoracic drainage within 24 hours
* controlled pain (below 3 points in the visual numeric scale, varying from zero to ten)

Exclusion Criteria:

* contraindication for use of noninvasive positive pressure in the airways, such as reduced level of consciousness (drowsiness, agitation or confusion), use of vasoactive drugs, complex arrhythmias, upper airway obstruction or trauma in the face, esophagus or upper airway, ineffective cough, inability to swallow, distended abdomen, nausea, vomiting, upper gastrointestinal bleeding
* previous application of any sort of lung expansion technique after thoracic drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Lung area | 20 seconds after pressure application

CONTACTS AND LOCATIONS:
Overall Officials: Adriana C Lunardi, PhD, Principal Investigator — Universidade Cidade de São Paulo

IPD SHARING:
Plan to Share IPD: No